CLINICAL TRIAL: NCT06603935
Title: Harnessing Digital Medicine Tools for Improving Allergic Rhinitis Control in the Primary Care Setting: Optimizing Management and Outcomes Via Technology
Brief Title: Harnessing Digital Medicine to Improve Allergic Rhinitis Management in Primary Care (DMAR)
Acronym: DMAR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: QHSLab, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: QHSLab 002-24
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Allergic Rhinitis; Sinusitis
Keywords: Allergic Rhinitis; Sinusitis; Digital Medicine; QHSLab; Allergy Management Evaluation; Allergic Rhinitis Intervention Steps; Digital Health Tools; Primary Care
MeSH Terms: conditions — Rhinitis, Allergic; Sinusitis | interventions — methylamphotericin B

STUDY DESIGN:
Intervention Model Description: This study utilizes a parallel assignment model. Participants are randomized into two groups: one group receives standard care (STC) for allergic rhinitis, and the other group receives both standard care and the use of the digital medicine tools, Allergy Management Evaluation (AME) and Allergic Rhinitis Intervention Steps (ARIS), provided through the QHSLab platform. The intervention group will receive continuous digital monitoring, personalized feedback, and treatment adjustments based on patient-reported outcomes. Both groups will be followed for 12 months with assessments at baseline, 3, 6, and 12 months to evaluate symptom severity, adherence, and healthcare utilization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (STC) group (No Intervention): Participants in this arm will receive the current standard of care for managing allergic rhinitis, which includes clinical evaluations, diagnosis, and treatments based on the healthcare provider's assessment. Treatment options may include medications such as intranasal corticosteroids, antihistamines, or decongestants, as typically prescribed for allergic rhinitis management. The standard care group will not have access to the digital tools provided in the experimental arm, but their care will follow established guidelines and practices for allergic rhinitis management.
- Standard Care plus Digital Tools (QHSLab with AME and ARIS) group (Experimental): Participants in this arm will receive the standard care for managing allergic rhinitis, which includes regular clinical evaluations and treatments as determined by their healthcare provider. In addition, they will be provided access to the QHSLab digital platform, which includes the Allergy Management Evaluation (AME) and Allergic Rhinitis Intervention Steps (ARIS) tools. These tools will offer continuous symptom monitoring, medication reminders, and personalized feedback based on patient-reported data. The intervention aims to improve symptom management, medication adherence, and quality of life over the 12-month follow-up period.
  Interventions: Other: QHSLab Digital Tools (AME and ARIS)

INTERVENTIONS:
Other: QHSLab Digital Tools (AME and ARIS) — Participants will use the QHSLab digital platform, which includes two tools: the Allergy Management Evaluation (AME) and the Allergic Rhinitis Intervention Steps (ARIS). The AME provides a comprehensive digital assessment for identifying and monitoring allergic rhinitis symptoms. The ARIS offers personalized feedback based on patient-reported outcomes and continuously adjusts treatment recommendations through an algorithm. These tools support better symptom management, adherence to medication, and overall improvement in quality of life.
  Arms: Standard Care plus Digital Tools (QHSLab with AME and ARIS) group

SUMMARY:
This study aims to evaluate the effectiveness of digital tools in managing allergic rhinitis (AR) in primary care settings. AR is a common condition that affects many people's quality of life. The study will test whether digital tools, such as the QHSLab platform, can help patients better control their symptoms, improve adherence to treatment, and enhance overall well-being. The trial will compare two groups: one using standard care and the other using both standard care and digital tools.

Participants will be monitored over 12 months, and the study will measure changes in symptom severity, treatment adherence, quality of life, and healthcare usage. The study will also gather feedback from patients and healthcare providers about their experience with the digital tools.

The digital tools used in this study are designed to help patients manage their AR more effectively by providing regular symptom assessments, medication reminders, and personalized feedback based on their health data.

This summary ensures the information is clear and straightforward for patients, families, and healthcare providers while maintaining compliance with IRB guidelines.

DETAILED DESCRIPTION:
This clinical trial is designed to assess the impact of integrating digital medicine tools on the management of allergic rhinitis (AR) in primary care settings. The study will compare outcomes between two groups: one receiving standard care (STC) and another receiving standard care plus digital tools from the QHSLab platform. The digital tools include the Allergy Management Evaluation (AME) and Allergic Rhinitis Intervention Steps (ARIS), both of which offer continuous monitoring, personalized feedback, and treatment optimization based on patient-reported outcomes.

The study is a prospective, randomized, controlled trial that will enroll 226 adult participants with uncontrolled allergic rhinitis, measured by the SNOT-22 score. Participants will be followed for 12 months, with data collection points at baseline, 3, 6, and 12 months. The study aims to evaluate:

Changes in symptom severity (SNOT-22 score). Medication adherence rates. Patient and provider satisfaction with the digital tools. Economic impact, including healthcare utilization and cost-effectiveness. Effects on mental health and quality of life. The study uses a mixed-methods approach, incorporating both quantitative measures and qualitative feedback through interviews with patients and healthcare providers to identify barriers and facilitators to adopting digital tools.

The QHSLab platform integrates seamlessly with current primary care workflows and includes tools for allergy management, offering insights based on patient interactions. The primary outcome is the reduction in symptom severity (SNOT-22 score), while secondary outcomes focus on patient adherence, healthcare use, satisfaction, and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* Clinically diagnosed with allergic rhinitis and/or sinusitis for at least 6 months.
* SNOT-22 score of ≥20, indicating uncontrolled allergic rhinitis.
* If Currently receiving treatment for allergic rhinitis and willing to continue treatment during the study.
* Able and willing to provide informed consent electronically and comply with the study procedures.

Exclusion Criteria:

* Individuals under 18 or over 65 years of age.
* Pregnant or breastfeeding women.
* Recent surgical treatment for nasal polyps (within the last 3 months).
* Patients with cystic fibrosis, purulent nasal infections, or any other disease likely to interfere with the study parameters.
* Individuals with severe or unstable concurrent diseases or psychological disorders that may compromise participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Allergic Rhinitis Symptom Severity (SNOT-22) | Baseline, 3 months, 6 months, 12 months
  This outcome measures the change in allergic rhinitis symptom severity using the SNOT-22 scale. Scores range from 0 to 110, with higher scores indicating worse symptoms and lower quality of life.
  unit: SNOT-22 score

SECONDARY OUTCOMES:
Change in Depression Symptoms (PHQ-9) | Baseline, 3 months, 6 months, 12 months
  This outcome measures the change in depressive symptoms using the Patient Health Questionnaire-9 (PHQ-9) scale. Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms and lower scores indicating fewer depressive symptoms and improved mental health.
  Unit: PHQ-9 score
Change in Anxiety Symptoms (GAD-7) | Baseline, 3 months, 6 months, 12 months
  This outcome measures the change in anxiety symptoms using the Generalized Anxiety Disorder-7 (GAD-7) scale. Scores range from 0 to 21, with higher scores indicating more severe anxiety and lower scores indicating fewer anxiety symptoms and improved mental health.
  Unit: GAD-7 score
Change in Quality of Life (Q-scale) | Baseline, 3 months, 6 months, 12 months
  This outcome measures the change in quality of life using the Q-scale, which assesses various aspects of a person's well-being, including relaxation, happiness, confidence, strain, pain, and satisfaction with family, work, and life. Scores range from 0 to 40, with higher scores indicating better quality of life and lower scores indicating higher risk and poorer quality of life.
  The scale is based on responses over the past 4 weeks, with items rated from "None of the time" to "All of the time." Unit: Q-scale score
Patient Satisfaction with Digital Tools (PDTS-10) | 3 months, 6 months, 12 months
  This 10-item scale measures patient satisfaction with the digital tools' ease of use and perceived effectiveness. Patients rate their agreement with statements on a 5-point Likert scale from 1 (Strongly Disagree) to 5 (Strongly Agree). Higher scores indicate higher satisfaction with the digital tools.
Provider Digital Tool Satisfaction Scale (PDTS-Provider) | Baseline, 3 months, 6 months, 12 months
  This scale measures healthcare providers' satisfaction with the ease of use and perceived effectiveness of the digital tools in improving patient care. Providers rate their agreement with statements on a 5-point Likert scale from 1 (Strongly Disagree) to 5 (Strongly Agree). Higher scores indicate higher satisfaction.
  PDTS-Provider score (Range: 10 to 50, higher scores indicate greater satisfaction)

CONTACTS AND LOCATIONS:
Locations (1):
- QHSLab, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data (IPD) will not be shared. The study will work with a compiled dataset that anonymizes and unifies all patient data, ensuring privacy and confidentiality

REFERENCES:
- [Background] Rizvi, S., et al. (2022). Allergies in Primary Care: A Study of the Allergy Management Evaluation Tool. Consultant, 62, e1-e8.